CLINICAL TRIAL: NCT04858880
Title: Personalized Radiotherapy for Biochemical Recurrence of Prostate Cancer After Prostatectomy: a Randomized Phase III Study.
Brief Title: Personalized Radiotherapy for Biochemical Recurrence of Prostate Cancer After Prostatectomy.
Acronym: PROPER2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-02
Record Dates: First submitted 2021-04-12; First posted 2021-04-26 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Prostate-Specific Antigen PSA; PSA; Radiation; Lymph node radiation; Prostate cancer recurrence; Randomized trial; Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continued salvage radiotherapy + lymph node irradiation (non responders) (Experimental): Continued salvage radiotherapy as initially planned (to 70.0 Gy/73.5 Gy in 35 fractions to the prostate bed/local recurrence if present) + the addition of lymph node irradiation (46 Gy/23 fractions) given in sequence. Total number of fractions: 35 + 8 = 43 with 15 of the lymph node irradiation fractions delivered concomitant with the prostate bed/local recurrence irradiation. These patients are classified as non responders according to weekly PSA measurements during the first 4 weeks of radiotherapy.
  Interventions: Radiation: Radiation to the prostate bed with or without addition of radiation of lymph node irradiation.
- Continued salvage radiotherapy (non responders) (Active Comparator): Continued salvage radiotherapy as initially planned (to 70.0 Gy/73.5 Gy in 35 fractions to the prostate bed/local recurrence if present). These patients are classified as non responders according to weekly PSA measurements during the first 4 weeks of radiotherapy.
  Interventions: Radiation: Radiation to the prostate bed with or without addition of radiation of lymph node irradiation.
- Continued salvage radiotherapy (responders) (No Intervention): Continued salvage radiotherapy as initially planned (to 70.0 Gy/73.5 Gy in 35 fractions to the prostate bed/local recurrence if present). These patients are classified as responders according to weekly PSA measurements during the first 4 weeks of radiotherapy, and are not followed according to the study protocol, follow up according to clinical practice.

INTERVENTIONS:
Radiation: Radiation to the prostate bed with or without addition of radiation of lymph node irradiation. — Radiation to the prostate bed with or without addition of radiation of lymph node irradiation (non responders). Patients with PSA response continues radiotherapy as initially planned, and are not followed according to the study protocol, only according to clinical practice.
  Arms: Continued salvage radiotherapy (non responders); Continued salvage radiotherapy + lymph node irradiation (non responders)

SUMMARY:
A randomized phase III trial to study the effect of adding lymph node irradiation in patients with poor prostate-specific antigen (PSA) response during salvage radiotherapy for biochemical recurrence (0.15 ≤ PSA <0.70 ng/ml) after prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy > 10 years
* Age ≥18 years.
* World Health Organization (WHO) performance status 0-1.
* Estimated life expectancy >10 years.
* Histological evidence of prostate cancer in the prostatectomy specimen
* Primary tumor, regional nodes, metastasis (TNM): any primary tumor (pT), pathologically node-negative (pN0), M0.
* Biochemical Recurrence (BCR) after prostatectomy, with 0.15 ≤ PSA <0.70 ng/ml.
* Patients must be able to comply with the protocol.
* Signed informed consent.
* Adequate laboratory findings (Haemoglobin (Hb) >90g/L, absolute neutrophil count >1.0x109/L, platelets >75x109/l, bilirubin <1.5x upper limit of normal (ULN), alanine aminotransferase (ALAT) <5x ULN and creatinine <1.5 ULN).

Exclusion Criteria:

* Metastases (regional lymph nodes or distant)* diagnosed with imaging.
* Prior or ongoing hormonal therapy (antiandrogens or gonadotropin releasing hormone).
* Prior radiotherapy to the pelvis.
* Prior malignancy other than prostate cancer and basalioma in the past five years.
* Clinically significant (i.e. active) cardiovascular disease e.g. myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) class III-IV congestive heart failure.
* Severe pulmonary disease.
* Any other serious or uncontrolled illness which in the opinion of the investigator makes it undesirable for the patient to enter the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only patients with prostate cancer are eligible.
Enrollment: 374 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS). | FFS after SRT, with failure defined as either biochemical or clinical recurrence (imaging or biopsy confirmed). FFS is calculated from the randomization date (arms A and B) until end of follow up (month 60 after
  Failure-free survival after salvage radiotherapy (SRT), with failure defined as either biochemical, defined as verified PSA level of ≥ 0.2 ng/ml above the post-radiotherapy PSA nadir value or clinical Recurrence, imaging or biopsy confirmed.

SECONDARY OUTCOMES:
Systemic treatment-free survival. | Is evaluated from the randomization date (arms A and B) until end of follow up (month 60 after end of radiotherapy).
  Arms A and B will be compared regarding systemic treatment-free survival.
Distant metastasis-free survival. | Is evaluated from the randomization date (arms A and B) until end of follow up (month 60 after end of radiotherapy).
  Arms A and B will be compared regarding distant metastasis-free survival. survival.
Prostate cancer specific survival. | Is evaluated from the randomization date (arms A and B) until end of follow up (month 60 after end of radiotherapy).
  Arms A and B will be compared regarding prostate cancer specific survival survival.
Overall survival. | Is evaluated from the randomization date (arms A and B) until end of follow up (month 60 after end of radiotherapy).
  Arms A and B will be compared regarding overall survival.
Numbers of patients with acute toxicity (≤ 3 months after end of salvage radiotherapy). | Up to 3 months after end of salvage radiotherapy.
  Toxicity that will be evaluated is presence of cystitis, bladder spasm, incontinence, urinary urgency, urinary retention, nausea, diarrhea, colitis, ileus, bloating, bowel obstruction, bowel perforation, gastrointestinal hemorrhage, rectal mucositis, erectile dysfunction, fatigue, lymphedema, pain, blood toxicity.
Numbers of patients with late toxicity (> 3 months to 5 years after end of salvage radiotherapy). | After 3 months after end of salvage therapy until end of follow up at month 60 after end of salvage therapy.
  Toxicity that will be evaluated is presence of cystitis, bladder spasm, incontinence, urinary urgency, urinary retention, nausea, diarrhea, colitis, ileus, bloating, bowel obstruction, bowel perforation, gastrointestinal hemorrhage, rectal mucositis, erectile dysfunction, fatigue, lymphedema, pain, blood toxicity.
Patients self-esteem of quality of life. | Quality of life evaluated using questionnaire by the European Organisation for Research and Treatment of Cancer (EORTC), questionnaire is QLQ-C30. Is done at baseline, at end of radiotherapy (43 days in Arm A, 35 days in Arm B), month 12, 24, and 60.
  Arms A and B will be compared regarding quality of life.
Patients self-esteem of quality of life. | Quality of life evaluated using questionnaire by the European Organisation for Research and Treatment of Cancer (EORTC), questionnaire is QLQ - PR25. Is done at baseline, at end of radiotherapy (43 days in Arm A, 35 days in Arm, month 12, 24, and 60.
  Arms A and B will be compared regarding quality of life.

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Jönköping County Hospital, Ryhov, Jönköping
  - Kalmar County Hospital, Kalmar
  - Lund University Hospital, Lund

IPD SHARING:
Plan to Share IPD: No